CLINICAL TRIAL: NCT04538313
Title: Early Clinical Trials on Evaluating the Tolerance, Safety and Efficacy of Autologous TILs in High-risk Recurrent Primary Hepatocellular Carcinoma
Brief Title: A Clinical Study in Patients With High-risk Recurrent Primary Hepatocellular Carcinoma Using Autologous TILs
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: CAR-T (Shanghai) Cell Biotechnology Co., Ltd. (Network)
Collaborators: Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: KT-2020-TIL001
Record Dates: First submitted 2020-08-26; First posted 2020-09-04 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-08

CONDITIONS: Hepatic Carcinoma
Keywords: TIL; HCC; clinical research
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- High dose group (Experimental): 10^10 TIL
  Interventions: Drug: Tumor infiltrating lymphocyte
- Low dose group (Experimental): 10^9 TIL
  Interventions: Drug: Tumor infiltrating lymphocyte
- Extension set (Experimental): The number of TIL is decided by dose escalation experiment.
  Interventions: Drug: Tumor infiltrating lymphocyte

INTERVENTIONS:
Drug: Tumor infiltrating lymphocyte — Tumor infiltrating lymphocytes were isolated from tumor tissues from tumor biopsy or operation. These TILs were cultured in human IL-2 medium for 4 to 5 weeks. 10e9 to 10e10 TILs were yielded. The phenotype, function and sterile were detected before these TILs infused patients.

SUMMARY:
Early clinical trials on evaluating the tolerance, safety and efficacy of autologous TILs in high-risk recurrent primary hepatocellular carcinoma

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years, gender unlimited;
2. Patients diagnosis of primary hepatocellular carcinoma by histopathology and/or cytology;
3. At the initial enrollment evaluation, patients were expected to accept radical resection of liver cancer and meet at least one of the following high-risk recurrence factors after surgery: ①There are 3 or more tumor lesions in the liver; ②The diameter of a single tumor lesion is >8cm; ③Existence macrovascular tumor thrombus; ④>5 MVI or MVI occurred in the distant paracancer tissues;
4. Before enrollment (after radical resection of liver cancer), imaging evaluation was performed to ensure that the tumor was completely removed (clear margin);
5. Must have at least 1 resectable lesion (diameter ≥2 cm);
6. ECOG score <2;
7. Child-Pugh score ≤7;
8. Hematology and organ function indicators should be met simultaneously: (1) White blood cell count ≥3.0E+9/ L, neutrophil count ≥1.5E+9/ L, platelet countPlatelet count ≥8.0E10/ L, hemoglobin ≥80g/L (2) Liver function: aspartate aminotransferase (AST)≤5 times normal value, alanine aminotransferase (ALT)≤5 times normal value, bilirubin ≤5 times normal value, serum albumin ≥28 g/L; (3) Renal function: creatinine (Cr)≤1.5 times normal limit, creatinine clearance ≥50 mL/min;
9. An estimated life expectancy of ≥3 months;
10. Participation in this clinical study voluntary, can cooperate with researchers to carry out research, and sign informed consent.

Exclusion Criteria:

1. Primary hepatocellular carcinoma (HCC) has recurred in the past, or has other types of liver cancer at the same time (such as intrahepatic cholangiocarcinoma, mixed type of liver cancer);
2. Have a history of high fever or severe infection within 2 weeks prior to pretreatment, or are expected to undergo systemic anti-infective therapy or systemic steroid therapy during this trial;
3. Hepatic encephalopathy occurred within 2 weeks before pretreatment;
4. Previous or screening with autoimmune liver disease;
5. Screening with moderate or higher peritoneal effusion;
6. Clear neurological/psychiatric symptoms are known to be associated with brain metastases and/or assessed by MMSE;
7. Anti-tumor therapy such as chemotherapeutic drugs, targeted drugs, radio frequency ablation or minimally invasive intervention was received within 4 weeks before pretreatment;
8. Have received or are expected to participate in this study within 4 weeks before pretreatment to receive TIL required focus radiotherapy, or tumor evaluation focus (target focus or non-target focus) radiotherapy, or radical radiotherapy;
9. Any toxic response resulting from previous anti-tumor treatment prior to pretreatment did not return to grade 1 or below (CTCAE5.0 version);
10. Previous history of organ / stem cell transplantation or expected to be involved in this trial for organ / stem cell transplantation;
11. Left ventricular ejection fraction (LVEF)<45% or New York Heart Association (NYHA)≥ grade 2;
12. Known or private HIV infection or syphilis infection;
13. The previous 3 years other system primary malignant tumor history (except skin basal cell carcinoma or cervical carcinoma in situ);
14. A known allergy to two or more non-homogeneous foods/drugs, or a known history of allergies to pre-treated drugs, including cyclophosphamide, fludarbin, interleukin;
15. Pregnant, lactating women or within one year of having a family plan;
16. Participated in other clinical trials within 3 months prior to screening;
17. Other circumstances that the researchers considered inappropriate to participate in the experiment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-08-26 (Actual); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
DLT | 24 months
  To evaluate the tolerability and safty of autologous TILs in high-risk recurrent primary hepatocellular carcinoma.
Progression-Free Survival | 24 months
  To evaluate the tolerability and safty of autologous TILs in high-risk recurrent primary hepatocellular carcinoma.

SECONDARY OUTCOMES:
Overall Survival Overall Survival | 24 months
  To evaluate the efficacy of autologous TILs in high-risk recurrent primary hepatocellular carcinoma.
EQ-5D score | 24 months
  To evaluate the efficacy of autologous TILs in high-risk recurrent primary hepatocellular carcinoma.

CONTACTS AND LOCATIONS:
Locations (1):
- Eastern Hepatobiliary Surgery Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided